CLINICAL TRIAL: NCT04021823
Title: Neurobiological Analyses Within the FORESEE III Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other); University Medical Center Freiburg (Other); University Hospital, Bonn (Other); University of Freiburg (Other)
Responsible Party: Principal Investigator, Thomas E. Schlaepfer, Prof. Dr., Professor Dr. Thomas E. Schläpfer, University Hospital Freiburg
Other Study IDs: 40418
Record Dates: First submitted 2019-06-24; First posted 2019-07-16 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; Neurobiological correlates of treatment resistant depression; Predictors of treatment response in DBS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DBS patients: Patients with treatment resistant major depression participating in the FORESEE III study.
- Healthy controls: Age- and sex-matched healthy controls undergoing analyses of neurodegenerative markers (neurofilament light protein) in blood and metabolomic analyses in blood and urine.

SUMMARY:
In this observational, non-invasive clinical study different neurobiological analyses will be performed in a group of patients with severe treatment resistant major depression participating in an efficacy study of deep brain stimulation of the superolateral branch of the medial forebrain bundle (slMFB) - FORESEE III.

DETAILED DESCRIPTION:
This study is a sub-project of the FORESEE III study (Controlled Randomized Clinical Trial to assess Efficacy of Deep Brain Stimulation (DBS) of the slMFB in Patients with Treatment Resistant Major Depression). The FORESEE III study itself is a randomized, sham-controlled, double blind (patient and observer blinded) clinical trial to assess the antidepressant effect of DBS compared to sham.

The aim of this sub-project is to analyze the time-course of biological correlates of treatment resistant major depression as well as neurobiological markers of treatment response to treatment with DBS in a well-characterized patient population during 12 month of DBS.

Specific neurobiological analyses include testing of

1. epigenetic markers (DNA methylation in candidate genes of depression and epigenome-wide association studies, EWAS)
2. markers of neuroinflammation (cytokines, neuropeptides and other immune factors)
3. micro RNAs and transcriptome signatures
4. markers of neurodegeneration (neurofilament light protein)
5. metabolomic analyses and
6. endocrinological parameters including glucose tolerance.

All markers will be tested in blood samples (and urine samples for metaboloic profiling) before neurosurgery as well as at several time points during DBS and sham condition intervals.

Additionally hemodynamic parameters will be analysed at test stimulation of the slMFB during neurosurgery.

The results will be correlated with clinical and other biological response parameters of the FORESEE III study and are hypothesized to indicate treatment response as well as allowing prediction of response to DBS. All neurobiological analyses will be linked in a tightly integrated and comprehensive translational approach.

Further, a volunteer group of healthy controls will be recruited and tested for blood-markers of neurodegeneration (neurofilament light protein, 4.) as well as metabolomic analyses in blood and urine (5.).

ELIGIBILITY:
DBS Patients:

Inclusion Criteria:

* All enrolled subjects of the Controlled Randomized Clinical Trial to assess Efficacy of Deep Brain Stimulation (DBS) of the slMFB in Patients with Treatment Resistant Major Depression (FORESEE III) may participate in this study.

Exclusion Criteria:

* Non-Caucasian (because of requirements for genetic/epigenetic analyses)
* Somatic diseases like diabetes, cancer and severe liver- and kidney-diseases

Healthy Controls:

Inclusion Criteria:

* All healthy volunteers without any clinically significant psychiatric or somatic symptoms are eligible.

Exclusion Criteria:

* Any clinically significant psychiatric symptoms
* Conditions like diabetes, cancer or severe liver- and kidney diseases
* Drug or alcohol abuse

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants are patients who participate in the FORESEE III study (NCT03653858) and have provided written informed consent to take part in this additional observational study. All patients suffering from severe, treatment-resistant depression, i.e. patients who have not sufficiently improved under established antidepressant therapies (such as psychotherapy, antidepressant drug therapy, and electroconvulsive therapy).
  As well as age- and sex-matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in DNA methylation patterns in plasma at 1 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 1 month of DBS (week 5 group A, week 21 group B)
  Epigenetic mechanisms such as DNA methylation crucially govern gene function and have been shown to be temporally dynamic and responsive to environmental stress. Epigenetic patterns in blood, saliva or other peripheral material have been suggested to partly reflect central epigenetic processes.
  DNA will by isolated and undergo bisulfite conversion. Using pyro- and direct sequencing, samples will be analyzed for DNA methylation in candidate genes of depression.
Change from baseline in DNA methylation patterns in plasma at 4 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 4 month of DBS (week 17 group A, week 33 group B)
  Epigenetic mechanisms such as DNA methylation crucially govern gene function and have been shown to be temporally dynamic and responsive to environmental stress. Epigenetic patterns in blood, saliva or other peripheral material have been suggested to partly reflect central epigenetic processes.
  DNA will by isolated and undergo bisulfite conversion. Using pyro- and direct sequencing, samples will be analyzed for DNA methylation in candidate genes of depression.
Change from baseline in DNA methylation patterns in plasma at 12 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 12 month of DBS (end of study both groups)
  Epigenetic mechanisms such as DNA methylation crucially govern gene function and have been shown to be temporally dynamic and responsive to environmental stress. Epigenetic patterns in blood, saliva or other peripheral material have been suggested to partly reflect central epigenetic processes.
  DNA will by isolated and undergo bisulfite conversion. Using pyro- and direct sequencing, samples will be analyzed for DNA methylation in candidate genes of depression.
Change from baseline in neuroinflammatory and neuropeptide patterns at 1 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 1 month of DBS (week 5 group A, week 21 group B)
  A new method of analysis (Proseek® Multiplex Inflammation, Olink Bioscience, Uppsala, Sweden) will be used to determine any change in patterns of relevant neuropeptides and inflammatory markers. This multiplex proximity extension assay (PEA) will simultaneously analyze 92 different proteins, including cytokines, neuropeptides and other immune factors.
Change from baseline in neuroinflammatory and neuropeptide patterns at 4 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 4 month of DBS (week 17 group A, week 33 group B)
  A new method of analysis (Proseek® Multiplex Inflammation, Olink Bioscience, Uppsala, Sweden) will be used to determine any change in patterns of relevant neuropeptides and inflammatory markers. This multiplex proximity extension assay (PEA) will simultaneously analyze 92 different proteins, including cytokines, neuropeptides and other immune factors.
Change from baseline in neuroinflammatory and neuropeptide patterns at 12 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 12 month of DBS (end of study both groups)
  A new method of analysis (Proseek® Multiplex Inflammation, Olink Bioscience, Uppsala, Sweden) will be used to determine any change in patterns of relevant neuropeptides and inflammatory markers. This multiplex proximity extension assay (PEA) will simultaneously analyze 92 different proteins, including cytokines, neuropeptides and other immune factors.
Change from baseline in transcriptome profiles at 1 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 1 month of DBS (week 5 group A, week 21 group B)
  A massive parallel next generation deep sequencing (NGS) technology will be used followed by bioinformatic network analysis to determine intraindividual changes in exosomal miR ( (miRs, 19-22 nt long non-coding RNAs) and transcriptome profiles.
Change from baseline in exosomal Micro-RNA (miR) expression levels and transcriptome profiles at 4 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 4 month of DBS (week 17 group A, week 33 group B)
  A massive parallel next generation deep sequencing (NGS) technology will be used followed by bioinformatic network analysis to determine intraindividual changes in exosomal miR ( (miRs, 19-22 nt long non-coding RNAs) and transcriptome profiles.
Change from baseline in exosomal Micro-RNA (miR) expression levels and transcriptome profiles at 12 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 12 month of DBS (end of study both groups)
  A massive parallel next generation deep sequencing (NGS) technology will be used followed by bioinformatic network analysis to determine intraindividual changes in exosomal miR ( (miRs, 19-22 nt long non-coding RNAs) and transcriptome profiles.
Change from baseline in plasma levels of Neurofilament light protein at 2 days before surgical device implantation | At baseline (up to 10 to 7 weeks before surgical device implantation) and at 2 days before surgical device implantation
  Neurofilament light protein is part of the neuroaxonal cytoskeleton and can be released into plasma following neuroaxonal damage. In plasma it will be measured by single-molecule array (SiMoA) assays.
Change from baseline in plasma levels of Neurofilament light protein at 1 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 1 month of DBS (week 5 group A, week 21 group B)
  Neurofilament light protein is part of the neuroaxonal cytoskeleton and can be released into plasma following neuroaxonal damage. In plasma it will be measured by single-molecule array (SiMoA) assays.
Change from baseline in plasma levels of Neurofilament light protein at 4 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 4 month of DBS (week 17 group A, week 33 group B)
  Neurofilament light protein is part of the neuroaxonal cytoskeleton and can be released into plasma following neuroaxonal damage. In plasma it will be measured by single-molecule array (SiMoA) assays.
Change from baseline in plasma levels of Neurofilament light protein at 12 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 12 month of DBS (end of study both groups)
  Neurofilament light protein is part of the neuroaxonal cytoskeleton and can be released into plasma following neuroaxonal damage. In plasma it will be measured by single-molecule array (SiMoA) assays.
Change from baseline in metabolite profiles in plasma and urine at 1 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 1 month of DBS (week 5 group A, week 21 group B)
  Metabolite profiles of plasma and urine samples will be analysed by chromatographic separation techniques, different mass spectrometric ionization modes and mass analyzers in order to assess molecular changes in the metabolome. The metabolomic methodologies may include fingerprinting, nontargeted, and targeted approaches, metabolic profiling and metabolic flux analysis.
Change from baseline in metabolite profiles in plasma and urine at 4 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 4 month of DBS (week 17 group A, week 33 group B)
  Metabolite profiles of plasma and urine samples will be analysed by chromatographic separation techniques, different mass spectrometric ionization modes and mass analyzers in order to assess molecular changes in the metabolome. The metabolomic methodologies may include fingerprinting, nontargeted, and targeted approaches, metabolic profiling and metabolic flux analysis.
Change from baseline in metabolite profiles in plasma and urine at 12 month of deep brain stimulation (DBS) | At baseline (up to 10 weeks before surgical device implantation) and at 12 month of DBS (end of study both groups)
  Metabolite profiles of plasma and urine samples will be analysed by chromatographic separation techniques, different mass spectrometric ionization modes and mass analyzers in order to assess molecular changes in the metabolome. The metabolomic methodologies may include fingerprinting, nontargeted, and targeted approaches, metabolic profiling and metabolic flux analysis.
Change from baseline in insuline resistance at week 41 | At baseline (up to 10 weeks before surgical device implantation) and at week 41 (both groups)
  An oral glucose tolerance test with blood measures of glucose, insulin and c-peptide at several time points during a period of 3 hours after oral intake of 75g glucose will be performed.
Change from baseline in systemic metabolic parameters at week 41 | At baseline (up to 10 weeks before surgical device implantation) and at week 41 (both groups)
  Different systemic metabolic parameters will be measured in blood.
Cardiac stroke volume (ml) | At test stimulation of the slMFB during neurosurgery
  Measured with ClearSight System, Edwards Lifesciences (allowing non-invasive and real-time continuous hemodynamic monitoring).
Non-invasive blood pressure (mmHG) | At test stimulation of the slMFB during neurosurgery
  Measured with ClearSight System, Edwards Lifesciences (allowing non-invasive and real-time continuous hemodynamic monitoring).
Cardiac stroke volume variation (%) | At teststimulation of the slMFB during neurosurgery
  Measured with ClearSight System, Edwards Lifesciences (allowing non-invasive and real-time continuous hemodynamic monitoring)
Systemic vascular resistance (mmHg⋅min⋅mL-1) | At test stimulation of the slMFB during neurosurgery
  Measured with ClearSight System, Edwards Lifesciences (allowing non-invasive and real-time continuous hemodynamic monitoring).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Schläpfer, Prof. Dr., Principal Investigator — University of Freiburg
Locations (1):
- University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Spanier S, Kilian HM, Meyer DM, Schlaepfer TE. Treatment resistance in major depression is correlated with increased plasma levels of neurofilament light protein reflecting axonal damage. Med Hypotheses. 2019 Jun;127:159-161. doi: 10.1016/j.mehy.2019.03.022. Epub 2019 Mar 23. PMID 31088642